CLINICAL TRIAL: NCT00600990
Title: Phase II Multicenter, Dose Ranging Study on the Safety and Antiemetic Efficacy of One Day Intraveous Dosing of GW597599 Administered With Ondansetron HCL in a Female Subjects Undergoing Surgical Procedures of High Emetogenic Risk
Brief Title: Study Of An NK-1 Anti-Emetic Medication For The Prevention Of Post-Operative Nausea And Vomiting In Female Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NKO101287
Record Dates: First submitted 2008-01-15; First posted 2008-01-25 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Postoperative Nausea and Vomiting; Nausea and Vomiting, Postoperative
Keywords: post-operative nausea and vomiting; PONV
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Vomiting | interventions — vestipitant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: GW597599

SUMMARY:
The purpose of this study is to determine the effectiveness of this medication in preventing nausea and vomiting in female patients at risk for post-operative nausea and vomiting (PONV).

DETAILED DESCRIPTION:
A Multicenter, Randomized, Double-blind, Double-dummy, Placebo-controlled, Parallel Group, Phase II Study to Evaluate the Safety, Efficacy, and Pharmacokinetics of Oral (25 mg) and Intravenous (3 mg and 18 mg) Formulations of the Neurokinin-1 Receptor Antagonist, GW597599, When Administered with Intravenous Ondansetron Hydrochloride for the Prevention of Post-operative Nausea and Vomiting and Post-discharge Nausea and Vomiting in Female Subjects with Known Risk Factors for PONV Who are Undergoing Surgical Procedures Associated with an Increased Emetogenic Risk

ELIGIBILITY:
Inclusion Criteria:

* known risk factors for PONV.
* Undergoing gynecological or gallbladder surgery.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 624 (Actual)
Dates: Start 2004-12; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
The number of subjects who achieve a complete antiemetic response during the first 24 hour evaluation period following the emergence from anesthesia.

SECONDARY OUTCOMES:
The number of subjects who achieve a complete antiemetic response during each subsequent 24 hour evaluation period (up to 120 hours) following the emergence from anesthesia.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (49):
- United States (16):
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Glendale, California
  - GSK Investigational Site, Laguna Hills, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Pasadena, California
  - GSK Investigational Site, Boca Raton, Florida
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Albany, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Spokane, Washington
- Australia (6):
  - GSK Investigational Site, St Leonards, New South Wales
  - GSK Investigational Site, Westmead, New South Wales
  - GSK Investigational Site, Carlton, Victoria
  - GSK Investigational Site, Melbourne, Victoria
  - GSK Investigational Site, Ringwood East, Victoria
  - GSK Investigational Site, Subiaco, Western Australia
- Belgium (3):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Leuven
- Canada (8):
  - GSK Investigational Site, Victoria, British Columbia
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Greater Sudbury, Ontario
  - GSK Investigational Site, Kingston, Ontario
  - GSK Investigational Site, Oshawa, Ontario
  - GSK Investigational Site, Charlottetown, Prince Edward Island
  - GSK Investigational Site, Chandler, Quebec
  - GSK Investigational Site, Regina, Saskatchewan
- GSK Investigational Site, Santiago, Región Metro de Santiago, Chile
- Czechia (4):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, Jihlava
  - GSK Investigational Site, Olomouc
  - GSK Investigational Site, Ostrava - Poruba
- Finland (2):
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Kuopio
- Netherlands (2):
  - GSK Investigational Site, Roosendaal
  - GSK Investigational Site, Rotterdam
- Poland (2):
  - GSK Investigational Site, Poznan
  - GSK Investigational Site, Warsaw
- South Africa (2):
  - GSK Investigational Site, Arcadia, Pretoria
  - GSK Investigational Site, Bloemfontein
- GSK Investigational Site, Istanbul, Turkey (Türkiye)
- United Kingdom (2):
  - GSK Investigational Site, Chelmsford, Essex
  - GSK Investigational Site, Northampton, Northamptonshire